CLINICAL TRIAL: NCT05506098
Title: Investigating STAT3 as a Driver of Pathology and Potential Therapeutic Target in Periodontitis
Brief Title: Investigating STAT3 as a Driver of Pathology in Periodontitis
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Nicolas Dutzan, Associate Professor, University of Chile
Other Study IDs: 11180389; FONDECYT 11180389 (Other Grant/Funding Number: AAgencia Nacional de Investigación y Desarrollo (ANID, Chilean Goverment))
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis
Keywords: periodontitis, STAT3
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gingival biopsies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: Subjects without periodontitis
  Interventions: Other: no intervention
- Periodontitis: Subjects with periodontitis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Periodontitis is a prevalent inflammatory condition that destroys tooth-supporting structures. This condition is associated with pro-inflammatory mediators that utilize STAT3 as an activator of specific genes related to inflammation and tissue destruction. STAT3 has not been studied in the context of periodontitis in humans. We propose that STAT3 is associated with periodontitis. This knowledge might help to further our understanding of periodontitis pathology

ELIGIBILITY:
Inclusion Criteria:

* 18-year-old, in good general health, and had no significant medical history.
* no history of diabetes or other diseases different than periodontitis.

Exclusion Criteria:

* Pregnancy and lactation
* Use of antibiotics, immunosuppressive agents, or probiotics within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male adults living in Santiago, Chile.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
STAT3 detection in gingival tissues | 1 day
  Detection of STAT3 in gingival tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
All data specified in the informed consent will be shared in publications
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: december 2022